

| HISTORY NUMBER: |
|-----------------|
| NAME: |
| Surname 1: |
| Surname 2: |
| Sex: |
| Data of hinth |

#### INFORMED CONSENT FOR GENERAL ANAESTHESIA - LOCOREGIONAL ANAESTHESIA

Anaesthesia is a procedure whose purpose is to perform a painless operation. In order to anaesthetise you, it is necessary to administer a series of cables and devices to monitor basic functions. There are numerous operations where it is convenient and necessary to perform general and locoregional anaesthesia at the same time (if this were your case, you would be informed of this).

The anaesthesiologist is in charge of controlling the entire process of anaesthesia from beginning to end and treating any complications that may arise.

Anaesthesia can involve some risks: the administration of serum and medicines, which are essential during anaesthesia, can produce exceptional allergic reactions, sometimes serious.

Scientific societies advise against the routine practice of allergy tests to anaesthetic drugs when there is no previous history of adverse reaction to them.

Furthermore, these tests are not risk-free and, even if the results are negative, the anaesthetics tested can produce adverse reactions during anaesthesia.

Furthermore, as a consequence of his clinical condition it may be necessary to transfuse him with blood. Each donation is analysed with the highest precision technique to detect certain diseases and infections (AIDS, hepatitis, etc.) transmitted by blood.

During a general anaesthetic, you will be asleep and generally relaxed. Tracheal intubation may be necessary. This tube is connected to a machine whose function is to oxygenate and provide adequate ventilation. Before or during tracheal intubation, part of the stomach contents may pass into the lung and cause significant respiratory disorders. TO REDUCE THIS RISK, IT IS NECESSARY TO FAST FOR AT LEAST 6 HOURS BEFORE SURGERY AND TO TAKE MEDICATION FOR THIS PURPOSE.

During regional anaesthesia there are also risks. On exceptional occasions, the drug can pass into the blood or nerve structures, producing serious complications such as a drop in blood pressure or convulsions, etc. These complications can be resolved but require the planned operation to be carried out under general anaesthesia.

If regional anaesthesia is not available or is not possible for technical reasons, general anaesthesia may be necessary.

After the administration of locoregional anaesthesia, there may be some discomfort, generally temporary, such as headache, backache, corkiness or tingling in the area.

| Your previous state of health may imply the existence of some personalised risks. The most significant | | |
|---|---|---|
| are; | | |
| I have been informed in an understandable manner of the usefulness, nature and risks of the above procedures, as well as of their alternatives. I am satisfied with the information I have received, being able to ask all the questions I | | |
| have thought fit, and having all 1 | | 2 |
| Patient | 's signature Doctor's signature | |
| Name of the local representative | ve in the event of the noticent's inch | ility to consent whether due to minerity legal |
| Name of the legal representative in the event of the patient's inability to consent, whether due to minority, legal incapacity or incompetence, indicating the nature of the intervention (father, mother, guardian, etc.) | | |
| Name | passport | |
| As theauthorizer of the above mentioned processes | | |
| DATE ToledoDEDE 20 | | |
| CANCELLATION OF CONS | | |
| _ | | ures, I freely and consciously express my refusal onsequences that may arise from this decision. |
| , | | • |
| Signature of patient Legal representative case | Signature of witness | Medical signature |
| | re in the event of the patient's inab | ility to consent, whether due to minority, legal |
| | icating the nature of the intervention | |
| Name | passport | |
| As theauthorizer of the above mentioned processes | | |
| D. (777 77 1.1) | | |
| DATE ToledoDE | DE 20 | |

# QUESTIONNAIRE AND ANSWERS FOR INTERVENTIONS OR COMPLEMENTARY FXAMINATIONS UNDER HYPNOSIS

## Taken from Montgomery 2000 and Virot & Bernard (146, 141)

#### What is hypnoanalgesia?

Hypnoanalgesia is a medical technique in which we use on the one hand the benefits of hypnosis to which we add analgesic drugs at low doses with fewer side effects, aiming at the patient's comfort and analgesia (without pain).

## What is hypnosis?

Hypnosis is a natural modified state of consciousness. It is possible to have experienced this state as a spontaneous hypnotic trance in our life without knowing it. Like driving our car automatically while our spirit escapes from our body for seconds.

In this way our brain allows us to live uncomfortable as well as pleasant moments. This natural spontaneous trance is neither long-lasting nor stable; for this reason with the help of a person trained in hypnosis using a technique, a voluntary hypnotic process can be created during medical care.

## Is it possible to use hypnosedation in all interventions?

All techniques have limitations. If this technique is proposed it is because it is intended to be so. Moreover, the patient must let himself go voluntarily, which implies motivation.

#### Is hypnosis dangerous?

Performed by a trained person and as an assistant within his competence is not dangerous. It is important to create the therapeutic alliance, obtaining the cooperation and trust of the patient.

# How does this process take place from the moment you arrive in the operating theatre?

On the day of the operation, he is initially in a room attached to the operating theatre and there he is received by the anaesthetist and nurse in the operating theatre. A check is made on your identity and medical history, and it is time to find out about your favourite place, your film, a pleasant walk, etc. No anaesthetic premedication is administered because scientific studies show that it is not useful. In the operating theatre, you are introduced to the rest of the team, the surgeon, the assistant and another nurse. You are comfortably seated on the operating table. Once installed, it is time to go mentally to that activity, a favourite place, fixing details.

With the help of a perfumed mask, you will start breathing a mixture of gases (O2/N2O) that will make you feel more relaxed at the same time. Products that produce analgesia are then injected. At this point, the surgeon places the sterile cloths on the area to be operated on and injects the local anaesthetic.

## Who will be watching during the intervention?

Throughout the surgery, the anaesthetist is responsible for monitoring the process and obtaining blood pressure, oxygen and heart rate measurements.

# What if at some point analgesia is insufficient?

Before the anaesthetic intervention, the patient and the anaesthetist agree to use some gesture in case of discomfort, such as lifting a finger, for example.

# Does this always work?

Collaboration between anaesthetist and patient is essential. There is absolute autonomy on the part of the patient. You cannot go against it, you can always change your mind.

## What if it doesn't work for me?

You will always be accompanied by an anaesthetist who can change the technique to general anaesthesia if necessary. You can change your mind from the anaesthesia consultation to the end of the operation.

## Is any special preparation required?

To make this experience easier, you could bring up the subject of the experience you are going to live in the operating theatre; memory of an unforgettable holiday, a bike trip, your favourite activity (gardening, painting...).